CLINICAL TRIAL: NCT05583006
Title: A Prospective Cohort Study of Tenofovir Alafenamide Switch Therapy in Chronic Hepatitis B Patients Who Are Unsatisfied to Entecavir Therapy
Brief Title: Tenofovir Alafenamide Switch Therapy in Chronic Hepatitis B
Status: Recruiting | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: Institute of Adherence to Medication (Unknown)
Responsible Party: Sponsor
Other Study IDs: CE22348B
Record Dates: First submitted 2022-10-14; First posted 2022-10-17 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Patient Satisfaction; Drug Adherence; Efficacy, Self; Safety Issues
MeSH Terms: conditions — Patient Satisfaction; Medication Adherence | interventions — tenofovir alafenamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: tenofovir alafenamide (TAF) — TAF switch therapy in CHB patients who are unsatisfied to ETV therapy.
  Other Names: Vemlidy

SUMMARY:
Chronic hepatitis B (CHB) patients may be unsatisfied to entecavir (ETV) therapy due to the inconvenience in drug taking, i.e., fasting for more than 2 hours and/or dose adjustment according to estimated glomerular filtration rate (eGFR). However, tenofovir alafenamide (TAF) has been approved to be highly effective and safe in patients with CHB, and is convenient in drug taking, i.e., once daily regardless food taking and renal function.Therefore,TAF can be a good option in CHB patients who are unsatisfied to ETV therapy. The aim of this prospective cohort study is to assess the improvement on satisfaction (including drug adherence) of TAF switch therapy in CHB patients who are unsatisfied to ETV therapy. In addition, with expected adherence improvement in TAF switch therapy, the efficacy of TAF switch therapy may be improved, and the efficacy benefits can be evaluated by the changes of some novel biomarkers, such as HBV core-related antigen (HBcrAg). The investigators therefore aim to conduct a prospective cohort study of TAF switch therapy for CHB patients who are unsatisfied to ETV therapy.

DETAILED DESCRIPTION:
Although nucleos(t)ide analogue (NA) therapy can effectively suppress HBV replication, the ideal therapeutic endpoints, including hepatitis B surface antigen(HBsAg) seroclearance, is difficult to achieve.(1) Therefore, chronic hepatitis B (CHB) patients often require long-term HBV suppression to achieve the therapeutic goals, with the adherence to long-term NA therapy being an important clinical issue.(2, 3) ETV is one of the standard treatments for CHB,(4, 5) but its absorption can be significantly reduced by food.(6) ETV users must take the pills two hours before or after meals, and the blood level of ETV may thus be affected if this recommendation is not fully followed.In addition, the metabolism of ETV is involved by renal excretion, therefore the dosage of ETV should be adjusted according to renal function.(7) For example, among patients in chronic kidney disease (CKD) stage 4, i.e.,eGRF15-29 ml/min/1.73m, the frequency of ETV taking should be reduced from once daily to every 72-96 hours, which may be forgettable and inconvenient to ETV users.However, the adherence of NA therapy is an essential part for long-term HBV suppression, and the efficacy of ETV therapy may be affected by the reduced adherence during long-term therapy.

Except ETV, TAF is also a HBV antiviral recommended by the current practice guidelines in the treatment of CHB, with a high potency in antiviral efficacy and low rate in virological resistance.(4, 5) In addition, TAF can be a 2nd-line rescue antiviral recommendation for HBV with resistance to ETV therapy.(4, 5) Moreover, because TAF is formulated to deliver the active metabolite to target cells more efficiently than tenofovir disoproxil fumarate (TDF) at a much lower dose, thereby reducing systemic exposure to tenofovir. In the randomized controlled trials,(8, 9) patients in the TAF arm had improved renal function and bone marrow density (BMD),as compared to patients in the TDF arm. Furthermore, in some retrospective studies, switching from ETV to TAF may present a superior efficacy in HBV DNA suppression and HBsAg level reduction,(10-13) and renal safety was comparable between the TAF switch group and the ETV continuation group.(10, 11) Interestingly, switching from ETV to TAF is associated with improvement of the medication adherence,(6) which may be particularly important to patients under long-term NA therapy.

In a small retrospective study conducted in Japan,(14) medication adherence and satisfaction were compared between before and after switch antiviral therapy in patients who switched to TAF from ETV (n = 15), and medication adherence was found to be significantly improved (P = 0.04). In a prospective study aimed to evaluate the changes of serum HBsAg levels during a 48-week period after switching ETV to TAF,(6) the degree of HBsAg reduction was higher during the TAF administration period than during the ETV administration period in patients without cirrhosis, with genotype B HBV, or with undetectable serum hepatitis B core-related antigen (HBcrAg).The HBV cccDNA-related biomarkers, such as quantitative HBsAg (qHBsAg) or HBcrAg, have been considered important outcome predictors.(15, 16) With expected adherence improvement in TAF switch therapy, the changes of above-mentioned biomarkers may be improved. The investigators therefore aim to conduct a prospective cohort study of TAF switch therapy for CHB patients who are unsatisfied to ETV therapy.

ELIGIBILITY:
Inclusion Criteria:

1. At least 20 years of age
2. Detectable serum HBsAg
3. Chronic HBV infection under ETV therapy
4. ETV users who are unsatisfied with the efficacy and/or feel inconvenient of ETV therapy
5. No contraindications for TAF switch therapy
6. HBV antiviral period expectancy for at least 1 year

Exclusion Criteria:

1. End stage renal disease (estimated glomerular filtration rate [eGRF]< 15 mL/min/1.73m2) without dialysis
2. Co-infected with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus
3. Any active malignancies
4. Under immunosuppressants
5. Known allergy to tenofovir-contained regimens

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective cohort study will enroll CHB patients who are unsatisfied to ETV therapy. The patient selection in this study is essentially based on a principle of shared decision making, and not only the physician decides whether to change the treatment. In the initial screening period, study subjects will be selected according to the inclusion and exclusion criteria, therefore only patients who complain the efficacy and/or inconvenience of ETV therapy (Inclusion criteria 4), will be invited to join this study. After discussing with the physician together, the study subjects must sign the inform consents before going into the next step (baseline condition evaluation).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate/ concentration of renal function markers | week 48
  The changes of eGFR, urine protein, urine beta 2-microglubulin, etc.
HBV viral load | week 48
The satisfaction (including drug adherence) to TAF switch therapy | week 48
  The changes of TSQM-9 questionnaire, MMAS-8 questionnaire

SECONDARY OUTCOMES:
Rate/ concentration of renal function markers | week 144
  The changes of eGFR, urine protein, urine beta 2-microglubulin, etc.
HBV viral load | week 144
The satisfaction (including drug adherence) to TAF switch therapy | week 144
  The changes of TSQM-9 questionnaire, MMAS-8 questionnaire
Concentration of biochemical markers | week 144
  bilirubin, AST, ALT

CONTACTS AND LOCATIONS:
Overall Officials: Teng-Yu Lee, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lok AS, Zoulim F, Dusheiko G, Ghany MG. Hepatitis B cure: From discovery to regulatory approval. J Hepatol. 2017 Oct;67(4):847-861. doi: 10.1016/j.jhep.2017.05.008. Epub 2017 Aug 1. PMID 28778687
- [Background] Sheppard-Law S, Zablotska-Manos I, Kermeen M, Holdaway S, Lee A, George J, Zekry A, Maher L. Factors associated with non-adherence to HBV antiviral therapy. Antivir Ther. 2018;23(5):425-433. doi: 10.3851/IMP3219. PMID 29355830
- [Background] Lee SS, Havens JP, Sayles HR, O'Neill JL, Podany AT, Swindells S, Scarsi KK, Bares SH. A pharmacist-led medication switch protocol in an academic HIV clinic: patient knowledge and satisfaction. BMC Infect Dis. 2018 Jul 6;18(1):310. doi: 10.1186/s12879-018-3226-2. PMID 29980192
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Uchida Y, Nakao M, Tsuji S, Uemura H, Kouyama JI, Naiki K, Motoya D, Sugawara K, Nakayama N, Imai Y, Tomiya T, Mochida S. Significance of switching of the nucleos(t)ide analog used to treat Japanese patients with chronic hepatitis B virus infection from entecavir to tenofovir alafenamide fumarate. J Med Virol. 2020 Mar;92(3):329-338. doi: 10.1002/jmv.25644. Epub 2019 Dec 9. PMID 31777965
- [Background] Yan JH, Bifano M, Olsen S, Smith RA, Zhang D, Grasela DM, LaCreta F. Entecavir pharmacokinetics, safety, and tolerability after multiple ascending doses in healthy subjects. J Clin Pharmacol. 2006 Nov;46(11):1250-8. doi: 10.1177/0091270006293304. PMID 17050790
- [Background] Chan HL, Fung S, Seto WK, Chuang WL, Chen CY, Kim HJ, Hui AJ, Janssen HL, Chowdhury A, Tsang TY, Mehta R, Gane E, Flaherty JF, Massetto B, Gaggar A, Kitrinos KM, Lin L, Subramanian GM, McHutchison JG, Lim YS, Acharya SK, Agarwal K; GS-US-320-0110 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of HBeAg-positive chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):185-195. doi: 10.1016/S2468-1253(16)30024-3. Epub 2016 Sep 22. PMID 28404091
- [Background] Buti M, Gane E, Seto WK, Chan HL, Chuang WL, Stepanova T, Hui AJ, Lim YS, Mehta R, Janssen HL, Acharya SK, Flaherty JF, Massetto B, Cathcart AL, Kim K, Gaggar A, Subramanian GM, McHutchison JG, Pan CQ, Brunetto M, Izumi N, Marcellin P; GS-US-320-0108 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of patients with HBeAg-negative chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):196-206. doi: 10.1016/S2468-1253(16)30107-8. Epub 2016 Sep 22. PMID 28404092
- [Background] Li ZB, Li L, Niu XX, Chen SH, Fu YM, Wang CY, Liu Y, Shao Q, Chen G, Ji D. Switching from entecavir to tenofovir alafenamide for chronic hepatitis B patients with low-level viraemia. Liver Int. 2021 Jun;41(6):1254-1264. doi: 10.1111/liv.14786. Epub 2021 Jan 19. PMID 33404182
- [Background] Hagiwara S, Nishida N, Ida H, Ueshima K, Minami Y, Takita M, Komeda Y, Kudo M. Switching from entecavir to tenofovir alafenamide versus maintaining entecavir for chronic hepatitis B. J Med Virol. 2019 Oct;91(10):1804-1810. doi: 10.1002/jmv.25515. Epub 2019 Jul 2. PMID 31199513
- [Background] Kumada T, Toyoda H, Tada T, Yasuda S, Miyake N, Tanaka J. Comparison of the impact of tenofovir alafenamide and entecavir on declines of hepatitis B surface antigen levels. Eur J Gastroenterol Hepatol. 2021 Feb 1;32(2):255-260. doi: 10.1097/MEG.0000000000001733. PMID 32282538
- [Background] Ogawa E, Nomura H, Nakamuta M, Furusyo N, Koyanagi T, Dohmen K, Ooho A, Satoh T, Kawano A, Kajiwara E, Takahashi K, Azuma K, Kato M, Shimoda S, Hayashi J; Kyushu University Liver Disease Study (KULDS) Group. Tenofovir alafenamide after switching from entecavir or nucleos(t)ide combination therapy for patients with chronic hepatitis B. Liver Int. 2020 Jul;40(7):1578-1589. doi: 10.1111/liv.14482. Epub 2020 Apr 30. PMID 32304611
- [Background] Tamaki N, Kurosaki M, Nakanishi H, Itakura J, Inada K, Kirino S, Yamashita K, Osawa L, Sekiguchi S, Hayakawa Y, Wang W, Okada M, Higuchi M, Takaura K, Maeyashiki C, Kaneko S, Yasui Y, Tsuchiya K, Takahashi Y, Izumi N. Comparison of medication adherence and satisfaction between entecavir and tenofovir alafenamide therapy in chronic hepatitis B. J Med Virol. 2020 Aug;92(8):1355-1358. doi: 10.1002/jmv.25692. Epub 2020 Feb 7. PMID 31994737
- [Background] Tseng TC, Liu CJ, Hsu CY, Hong CM, Su TH, Yang WT, Chen CL, Yang HC, Huang YT, Fang-Tzu Kuo S, Liu CH, Chen PJ, Chen DS, Kao JH. High Level of Hepatitis B Core-Related Antigen Associated With Increased Risk of Hepatocellular Carcinoma in Patients With Chronic HBV Infection of Intermediate Viral Load. Gastroenterology. 2019 Dec;157(6):1518-1529.e3. doi: 10.1053/j.gastro.2019.08.028. Epub 2019 Aug 27. PMID 31470004
- [Background] Tseng TC, Liu CJ, Yang WT, Hsu CY, Hong CM, Su TH, Tsai CH, Chen CL, Yang HC, Liu CH, Chen HH, Chen PJ, Kao JH. Serum hepatitis B core-related antigen level stratifies risk of disease progression in chronic hepatitis B patients with intermediate viral load. Aliment Pharmacol Ther. 2021 Apr;53(8):908-918. doi: 10.1111/apt.16266. Epub 2021 Jan 19. PMID 33465271
- [Background] Bharmal M, Payne K, Atkinson MJ, Desrosiers MP, Morisky DE, Gemmen E. Validation of an abbreviated Treatment Satisfaction Questionnaire for Medication (TSQM-9) among patients on antihypertensive medications. Health Qual Life Outcomes. 2009 Apr 27;7:36. doi: 10.1186/1477-7525-7-36. PMID 19397800